CLINICAL TRIAL: NCT03999957
Title: CALLiNGS Protocol: Care Across Locations Longitudinally in Navigation of Goals and Symptoms (Interdisciplinary Pediatric Telepalliative Consultations for Hospice Teams)
Brief Title: CALLiNGS Protocol: Care Across Locations Longitudinally in Navigation of Goals and Symptoms
Acronym: CALLiNGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0454-18-EP
Record Dates: First submitted 2019-06-18; First posted 2019-06-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Palliative Care
Keywords: hospice; pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Other): Telehealth conferencing
  Interventions: Other: Telehealth web conferencing

INTERVENTIONS:
Other: Telehealth web conferencing — Pediatric patient specific case discussions for enrolled pediatric patients at hospice staff interdisciplinary team meeting every 15 days for 60 min sessions via telehealth

SUMMARY:
The study intends to explore feasibility, acceptability, and quality of life outcomes from using web-conferencing technology to connect a hospital-based interdisciplinary pediatric palliative care with statewide field-based hospice teams during interdisciplinary meetings at a minimum of every 15 calendar days for a maximum of six months per enrollee.

DETAILED DESCRIPTION:
The Central Hypothesis is that telepalliative care has the potential to improve the quality of care delivered to pediatric palliative care patients in a rural state by connecting local care providers with palliative care interdisciplinary subspecialists at an academic health center to facilitate improved symptom burden which translates into enhanced quality of life for the pediatric patient and family members, increased confidence and comfort of local providers, and ultimately the creation of a unified and cross-setting shared care model.

Aim 1. To investigate the symptom burden for pediatric patients and the quality of life impact for pediatric patients and their families through an interdisciplinary pediatric telepalliative consultation service partnered with local hospice providers with an interface at a minimum of every 15 day intervals.

Aim 2. To evaluate the self-efficacy, knowledge, and self-perceived adequacy of local hospice providers in caring for pediatric patients before and after interdisciplinary pediatric telepalliative consultation service partnership with these local hospice providers.

Aim 3. To explore the acceptability of teleconferencing services as a form of pediatric palliative care mentorship for local hospice teams caring for children and adolescents.

Expected Outcomes Based on geography and shortage of pediatric palliative subspecialists in Nebraska, the current model of hospice services is one in which pediatric patients are managed by local adult-based hospice teams after discharge from the pediatric hospital (34 such in the past 16 months). Sixty percent of academic pediatricians in Nebraska who served as primary providers for consecutive pediatric home discharge patients self-reported feeling "very deficient" to "deficient" when asked about competence after supporting terminal patients and families in care at home (n=12).1 The knowledge gap and discomfort in managing children with complex symptom burden is magnified further for family practice or internal medicine teams serving in hospice roles for children in rural communities. Through a new telepalliative technology platform, this study fosters collaboration and communication to improve the quality of care for pediatric patients receiving hospice care in rural states. This model implements human interaction through technology to challenge the existing paradigm of silo-based care of pediatric palliative care patients. With roll-out of this intervention, we anticipate increase in pediatric hospice utilization (decreased in-hospital deaths). If feasible this model could transform the pediatric hospice care delivery in the state of Nebraska with expanded opportunity for application in settings with similar subspecialty provider shortages.

ELIGIBILITY:
Inclusion Criteria:

* age birth to 18 years.
* Enrolling on home hospice services within the state of Nebraska at time of discharge from the hospital.

Exclusion Criteria:

* Age older than age 18 years
* Does not speak English
* Not enrolling in home hospice services within the state of Nebraska at time of discharge from the hospital

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
To investigate quality of life trend over time for pediatric participants and their families | Every 15 days for a total of 3 months
  Using patient-reported & proxy reported pediatric quality of life metrics longitudinally with pediatric quality of life scale completion by patient & proxy every 15 days for a total of 3 months. The PedsQL™ 4.0 Generic Core Parent Report measures proxy perception on a child's quality of life. The 21-item PedsQL™ 4.0 Generic Core consists of the following dimensions: physical functioning, emotional functioning, social functioning, and school functioning.
  Participants are asked how much of a problem each survey item has been during the past one month. A 5-point response scale is utilized (0 = never; 4 = almost always).
  On the PedsQL™ 4.0 Generic Core Parent Report items are so that higher scores indicate better Health-Related Quality of Life. To reverse score, the 0-4 scale items are translated to 0-100 as follows: 0=100, 1=75, 2=50, 3=25, 4=0. To create the Total Scale Score, the mean is computed as the sum of all the items over the number of items answered on all the Scales.
To evaluate the change in perception of adult-trained hospice providers about caring for pediatric patients on hospice | Day 1 of study and at Month 3
  2 qualitative interview questions asked on Day 1 with the same 2 questions asked again on Month 3. The questions are as follows: a) Please describe your experience caring for a pediatric patient. b) Please describe your experience with telepalliative use.
To monitor change in telehealth technology acceptance over two week time | Day 1 and again on Day 14
  TAM-2 Scale (Technology Acceptance Model) completed on Day 1 and Day 14= two time points. The Technology Acceptance Model (TAM2) is a 15-item questionnaire that measures acceptability of a technology modality. The Technology Acceptance Model (TAM2) was developed to gauge individuals' intentions and behaviors for technology usage. TAM2 topics include perceived usefulness, ease of use and learnability, interface quality, interaction quality, reliability, satisfaction, and future use. Responses are on a five-point Likert scale (from 1= "highly disagree" to answer 5="highly agree"). Responses are tallied for a total score with a higher score correlating with a higher level of approval/acceptance of the technology modality.

CONTACTS AND LOCATIONS:
Overall Officials: Meaghann S Weaver, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska

REFERENCES:
- [Background] Weaver MS, Reeve BB, Baker JN, Martens CE, McFatrich M, Mowbray C, Palma D, Sung L, Tomlinson D, Withycombe J, Hinds P. Concept-elicitation phase for the development of the pediatric patient-reported outcome version of the Common Terminology Criteria for Adverse Events. Cancer. 2016 Jan 1;122(1):141-8. doi: 10.1002/cncr.29702. Epub 2015 Sep 30. PMID 26421973
- [Background] Rosenberg AR, Orellana L, Ullrich C, Kang T, Geyer JR, Feudtner C, Dussel V, Wolfe J. Quality of Life in Children With Advanced Cancer: A Report From the PediQUEST Study. J Pain Symptom Manage. 2016 Aug;52(2):243-53. doi: 10.1016/j.jpainsymman.2016.04.002. Epub 2016 May 21. PMID 27220948
- [Background] Rodgers C, Hooke MC, Ward J, Linder LA. Symptom Clusters in Children and Adolescents with Cancer. Semin Oncol Nurs. 2016 Nov;32(4):394-404. doi: 10.1016/j.soncn.2016.08.005. Epub 2016 Oct 21. PMID 27776834
- [Background] Rodgers CC, Hooke MC, Hockenberry MJ. Symptom clusters in children. Curr Opin Support Palliat Care. 2013 Mar;7(1):67-72. doi: 10.1097/SPC.0b013e32835ad551. PMID 23108342
- [Background] Wang J, Jacobs S, Dewalt DA, Stern E, Gross H, Hinds PS. A Longitudinal Study of PROMIS Pediatric Symptom Clusters in Children Undergoing Chemotherapy. J Pain Symptom Manage. 2018 Feb;55(2):359-367. doi: 10.1016/j.jpainsymman.2017.08.021. Epub 2017 Sep 1. PMID 28865867
- [Background] Lee SE, Vincent C, Finnegan L. An Analysis and Evaluation of the Theory of Unpleasant Symptoms. ANS Adv Nurs Sci. 2017 Jan/Mar;40(1):E16-E39. doi: 10.1097/ANS.0000000000000141. PMID 27525959
- [Background] Brown SJ. Integrating and synthesizing work on middle-range theories. ANS Adv Nurs Sci. 1996 Jun;18(4):vi-vii. doi: 10.1097/00012272-199606000-00001. No abstract available. PMID 8790684
- [Background] Cody WK. Middle-range theories: do they foster the development of nursing science? Nurs Sci Q. 1999 Jan;12(1):9-14. doi: 10.1177/089431849901200106. No abstract available. PMID 11847659
- [Background] Lenz ER, Suppe F, Gift AG, Pugh LC, Milligan RA. Collaborative development of middle-range nursing theories: toward a theory of unpleasant symptoms. ANS Adv Nurs Sci. 1995 Mar;17(3):1-13. doi: 10.1097/00012272-199503000-00003. PMID 7778887
- [Background] Pilkington FB. Development of middle-range theories. Nurs Sci Q. 2006 Jul;19(3):277-80. No abstract available. PMID 16838432
- [Background] Dirksen SR, Belyea MJ, Epstein DR. Fatigue-based subgroups of breast cancer survivors with insomnia. Cancer Nurs. 2009 Sep-Oct;32(5):404-11. doi: 10.1097/NCC.0b013e3181a5d05e. PMID 19661794
- [Background] Hoffman AJ, von Eye A, Gift AG, Given BA, Given CW, Rothert M. Testing a theoretical model of perceived self-efficacy for cancer-related fatigue self-management and optimal physical functional status. Nurs Res. 2009 Jan-Feb;58(1):32-41. doi: 10.1097/NNR.0b013e3181903d7b. PMID 19092553
- [Background] Hsu MC, Tu CH. Improving quality-of-life outcomes for patients with cancer through mediating effects of depressive symptoms and functional status: a three-path mediation model. J Clin Nurs. 2014 Sep;23(17-18):2461-72. doi: 10.1111/jocn.12399. Epub 2013 Sep 21. PMID 24112217

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03999957/Prot_SAP_000.pdf